CLINICAL TRIAL: NCT01216982
Title: Effects of Omega-3 EPA/DHA for Soldiers at Risk for Mood Disorders: A Mood Resilience Trial
Brief Title: Effects of Omega-3 EPA/DHA for Soldiers at Risk for Mood Disorders
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: United States Department of Defense (U.S. Federal Agency)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Daniel T. Johnston, MD, MPH, LTC, US Army MC,, 1st CAB, US ARMY
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: M-10023
Record Dates: First submitted 2010-10-06; First posted 2010-10-07 (Estimated); Last update posted 2011-03-09 (Estimated); Status verified 2011-03

CONDITIONS: Mood Disorders; Depression; Combat Disorders; Stress Disorders
Keywords: Mood Disorders; Depression; Combat Disorders; Stress Disorders; Fatty Acids, Omega-3; Military Personnel; Docosahexaenoic Acids/*therapeutic use; Eicosapentaenoic Acid/*therapeutic use
MeSH Terms: conditions — Mood Disorders; Depression; Combat Disorders; Stress Disorders, Traumatic | interventions — Omacor; Corn Oil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Lovaza, omega-3 fatty acid ethyl ester (Active Comparator)
  Interventions: Drug: Lovaza, omega-3 fatty acid ethyl ester
- Placebo (Placebo Comparator): one gram corn oil in a soft gelatin capsule
  Interventions: Drug: Placebo, visually identical to Lovaza

INTERVENTIONS:
Drug: Lovaza, omega-3 fatty acid ethyl ester — Three 1g capsules/day for three months; this corresponds to a total of 2520mg EPA+DHA/day
  Other Names: LOVAZA 1g Soft Gelatin Capsules NDC NO. 65726-425-15; Omega-3-Acid Ethyl Esters
  Arms: Lovaza, omega-3 fatty acid ethyl ester
Drug: Placebo, visually identical to Lovaza — Three 1g corn oil capsules/day for three months
  Other Names: Corn oil
  Arms: Placebo

SUMMARY:
Stress-related disorders are among the most prevalent and expensive medical consequences of participation in military operations. Omega-3 fatty acids EPA/DHA derived from fish oil are known to benefit both neuronal development in the young, and cognition and mood in various populations.

It is possible that soldiers receiving Omega-3 EPA/DHA will exhibit significantly higher cognitive performance, better affect/mood state, and less combat stress symptomatology compared to the placebo after 12 weeks of supplementation. A goal would be to reduce the prevalence of combat stress injuries in military personnel.

ELIGIBILITY:
Inclusion Criteria:

* US Army deployed personnel
* score on a mood questionnaire

Exclusion Criteria:

* currently consume omega-3 fish oil supplements
* are currently taking antidepressant or other medications for psychiatric purposes
* pregnant
* known fish or shellfish allergy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 256 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-02 (Actual); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
primary psychometric assessment battery | 3 months
  Specific components include:
  Zung Depression Scale (ZDS) Zung Anxiety Scale (ZAS) Pittsburgh Sleep Quality Index (PSQI) Epworth Sleepiness Scale (ESS)
omega-3 fatty acid status | 3 months
  finger-prick blood spot is collected for determination of fatty acid composition and profile.

SECONDARY OUTCOMES:
secondary psychometric assessment battery | 3 months
  This battery will generate index scores in the area of:
  Memory, Psychomotor Speed, Reaction Time, Cognitive Flexibility, and Complex Attention. It will also include the Alcohol Use Identification Test (AUdIT). Military-specific components include Post-Deployment Health Assessment (PDHA), Neurobehavioral Symptom Inventory (NSI), Combat Exposure Scale (CES), and parts of the Deployment Risk and Resilience Inventory (edited).

CONTACTS AND LOCATIONS:
Overall Officials: Daniel T Johnston, MD, MPH, Principal Investigator — United States Department of Defense
Locations (1):
- US Military Base, Camp Taji, Iraq